CLINICAL TRIAL: NCT03450083
Title: Benralizumab Effect on Severe Chronic Rhinosinusitis With Eosinophilic Polyposis: A Phase II Randomized Placebo Controlled Trial
Brief Title: Benralizumab Effect on Severe Chronic Rhinosinusitis With Eosinophilic Polyposis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00112910
Record Dates: First submitted 2017-08-17; First posted 2018-03-01 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Nasal Polyps; Eosinophilia
MeSH Terms: conditions — Disease; Nasal Polyps; Eosinophilia | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Benralizumab treatment group (Active Comparator): Benralizumab Active treatment group delivered subcutaneously
  Interventions: Drug: Benralizumab
- Placebo group (Placebo Comparator): Placebo treatment group delivered subcutaneously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benralizumab — 30mg Benralizumab will be delivered subcutaneously
  Other Names: Fasenra
  Arms: Benralizumab treatment group
Drug: Placebo — Subcutaneous placebo injection
  Arms: Placebo group

SUMMARY:
Benralizumab will be used in a placebo controlled randomized study to treat severe chronic rhinosinusitis with nasal polyps

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) has a prevalence of more than 10% in the United States and Europe and is associated with several co-morbidities including asthma, acute infection, and obstructive sleep apnea. There are principally two forms of CRS namely with and without nasal polyps. CRS with nasal polyps (CRSwNP) in particular can be a severe and debilitating disease resulting in significant morbidity, complete anosmia, headaches, missed work, and hospitalizations. Not uncommonly, patients require chronic oral corticosteroids, multiple courses of antibiotics, and repeated surgical polypectomies to control participants' disease. Total health care expenditure for CRS (which includes both with and without polyps) is more than $60 billion annually in the United States accounting for as much as 5% of the total US health care budget. Annual direct and indirect costs to treat CRS in Europe is estimated to be similar to this amount but data is limited.

For CRSwNP patients suffering with severe and recurrent nasal polyps there are few treatment options. High dose topical nasal steroids and repeated surgical procedures do not halt progression in many patients. Allergen immunotherapy is often non-curative in this population. Similarly, due to the fact that CRSwNP is not exclusively an Immunoglobulin E (IgE) driven process, omalizumab was shown to have mixed benefit in this population. Likewise, omalizumab resulted in no reduction in polyp size among patients with Aspirin Exacerbated Respiratory Disease (AERD).

More typically chronic nasal polyp disease is an eosinophil mediated process. Patients with demonstrated elevations in serum and mucosal eosinophils tend to have more severe disease and higher nasal polyp recurrence rates. Clinical researchers have begun to recognize this connection. A recent Phase II study in Europe showed a reduction in polyp burden using mepolizumab anti-Interleukin (IL) 5 monoclonal antibody. Benralizumab which targets IL-5 receptor signaling has been shown to have powerful apoptotic effects on eosinophils and may likely prove to be even more efficacious. Because of its unique mechanism of action, benralizumab may have a profound impact on reducing mucosal eosinophils resulting in great benefit to patients suffering with severe nasal polyps refractory to standard treatment.

Benralizumab has been shown to be efficacious treating severe asthmatics with eosinophilia. The unique mechanism of action of benralizumab targets the IL-5 receptor leading to degradation of signaling and apoptosis. This direct effect on eosinophils leads to reduction of proinflammatory processes in the asthmatic airways among those with elevated eosinophil counts. While many subjects with allergic asthma do indeed have concomitant local and systemic elevations in eosinophils, the primary driver of inflammation in allergic asthmatics is IgE and IL-4. Allergen immunotherapy and anti-IgE therapy (omalizumab) has long been known to be effective in these atopic individuals. However, a significant portion of non-asthmatics respond poorly to these IgE targeted therapies.

In a similar manner, chronic rhinosinusitis with nasal polyps (CRSwNP) is a disease often associated with atopy and propagated by IgE/IL-4 mediated inflammation. However, more than 50% of patients with CRSwNP have no evidence of allergen sensitivity. Nasal and sinus inflammation in these non-atopic individuals is often characterized by IL-5 upregulation, eosinophilia, leukotrienes, and more severe polyps. These individuals tend to have more aggressive disease requiring frequent surgeries, high dose intranasal budesonide irrigation, and oral steroids yet the polyps more often than not are persistent and may return post surgery. In a subset of patients, concomitant aspirin sensitivity can be managed with aspirin desensitization, however this approach is not always effective and can also be cumbersome. A more universal and potentially more efficient approach to treating severe polyps is to target eosinophils directly using a monoclonal antibody. Previous reports have shown some benefit targeting IL-5 ligand itself with mepolizumab but the potential benefit of directly eliminating eosinophils by shutting down cellular signaling with benralizumab would be expected to have a more dramatic effect and needs to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75
* Severe bilateral nasal polyps with average endoscopic score of at least 5
* Blood eosinophil count of at least 300/ul at screening
* At least 1000mg prednisone (or equivalent) over the previous 12 months to control symptoms
* At least one prior nasal surgical polypectomy
* Informed Consent: Able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. Subjects must be able to read, comprehend, and write at a level sufficient to complete study related materials.
* Female subjects: Women of childbearing potential (WOCBP) must use an effective form of birth control (confirmed by the Investigator). Effective forms of birth control include: true sexual abstinence, a vasectomized sexual partner, Implanon, female sterilization by tubal occlusion, any effective Intra-uterine device (IUD) intrauterine device/ levonogestrel Intrauterine system (IUS), Depo-Provera(tm) injections, oral contraceptive, and Evra Patch(tm) or Nuvaring(tm). WOCBP must agree to use effective method of birth control, as defined above, from enrolment, throughout the study duration and within 16 weeks after last dose of IP, and have negative serum pregnancy test result on Visit 0.
* Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for 12 months prior to the planned date of visit -1 without an alternative medical cause. The following age-specific requirements apply:
* Women <50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
* Women ≥50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.
* All male subjects who are sexually active must agree to use an acceptable method of contraception (condom with or without spermicide, vasectomy) from Visit 0 until 16 weeks after their last dose.

Exclusion Criteria:

* Immunosuppression other than oral steroids in the past 3 months
* Allergen immunotherapy build up phase in the past 3 months
* Symptomatic or untreated life threatening cardiopulmonary disorders
* Subjects who are febrile (≥38°C; ≥100.4°F);
* History of cancer: Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to the date informed consent, and assent when applicable was obtained. Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to the date informed consent, and assent when applicable, was obtained.
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.
* Pregnant or nursing
* If female and of child-bearing potential, positive pregnancy test or failure to adhere to acceptable method of contraception (with <1% failure rate) during the study and for four months after the study.
* Receipt of any investigational non biologic within 30 days or 5 half-lives prior to visit 0, whichever is longer.
* A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
* Any other medical illness that precludes study involvement
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to be enrolled.
* Patients who are currently receiving or have previously received benralizumab or any other type of anti-interleukin therapy (i.e. mepolizumab, reslizumab, lebrikizumab etc.) within the last 4 months or 5 half-lives whichever is longer.
* History of anaphylaxis to any biologic therapy or vaccine.
* Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent is obtained.
* Receipt of live attenuated vaccines within 30 days of starting the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jody Tversky, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geng B, Dilley M, Anterasian C. Biologic Therapies for Allergic Rhinitis and Nasal Polyposis. Curr Allergy Asthma Rep. 2021 Jun 10;21(6):36. doi: 10.1007/s11882-021-01013-y. PMID 34110505
- [Derived] Tversky J, Lane AP, Azar A. Benralizumab effect on severe chronic rhinosinusitis with nasal polyps (CRSwNP): A randomized double-blind placebo-controlled trial. Clin Exp Allergy. 2021 Jun;51(6):836-844. doi: 10.1111/cea.13852. Epub 2021 Feb 27. PMID 33595845

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 participants signed Informed Consent; 2 participants did not meet inclusion criteria and 7 participants decided to not continue with study activities prior to receiving any intervention.
Period: Overall Study
Arm/Group | Benralizumab Treatment Group | Placebo Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 49.8 [33 to 70] | 50.8 [35 to 67] | 50.3 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Nasal Polyp Score
Description: Change in endoscopic nasal polyp score after 6 months of treatment. Nasal Polyp Score (NPS): the change in mean score from Screen visit (Week 5) bilateral endoscopic nasal polyp score as compared to score at end of treatment (Week 25). Higher scores indicate increase in number of polyps and/or polyp size. The score is the sum of the right and left nostril scores, as evaluated by nasal endoscopy.
  NPS score key: 0 = No visible polyps; 1 = Small amount of polypoid disease confined within the middle meatus; 2 = Multiple polyps occupying the middle meatus; 3 = Polyps extending beyond the middle meatus; 4 = Polyps completely obstructing the nasal cavity.
  Reported data is a difference in the NPS between Week 25 and Week 5.
Time Frame: Week 5 and Week 25
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
score on a scale | .9 [0 to 3] | .3 [-1 to 2]

2. Secondary Outcome: Change in Nasal Polyp Size as Assessed by the Lund Mackay Score
Description: Computed Tomography (CT) scan of the sinus was performed at screening (Week 5) and then again at the end of treatment (Week 25). Sinus CT images were obtained to determine the Lund Mackay Score (LMS), a widely used method for radiologic staging of nasal polyposis. The mean change in the LMS was determined by comparing the scores from Week 5 to Week 25. Each sinus group is graded between 0 and 2 (0: no abnormality; 1: partial opacification; 2: total opacification). The ostiomeatal complex is scored as "0" not obstructed) or "2" (obstructed). Overall score range of 0-24. Higher scores indicate progression of nasal polyposis disease.
  Reported data is a difference in the LMS between Week 25 and Week 5.
Time Frame: Week 5 and Week 25
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
score on a scale | -4.2 (1.1) | -1.6 (1.2)

3. Secondary Outcome: Change in Symptom Severity Score as Assessed by the Sino-nasal Outcome Test
Description: The Sino-nasal Outcome Test (SNOT-22) is a condition-specific health-related quality of life assessment that captures patient-reported physical problems, functional limitations, and emotional consequences of sinonasal conditions for the 2 weeks prior to completing the test. Participants completed the SNOT-22 at treatment Week 0 and at Treatment Week 20. Patients rated their symptom severity and symptom impact over the previous 2 weeks using a 6-point scale (0- No Problem to 5- Problem as bad as it can be). The total score is the sum of individual item scores and has a range from 0 to 110. Higher scores indicate more severe symptoms. Outcome measure data shows change in SNOT-22 scores between treatment Week 20 and Week 0.
Time Frame: Treatment Week 0 and Week 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
score on a scale | -19.2 (2.6) | -14.6 (20.1)

4. Secondary Outcome: Change in The University of Pennsylvania Smell Identification Test Score
Description: The University of Pennsylvania Smell Identification Test (UPSIT) is a quantitative test of olfactory function that uses microencapsulated odorants that are released by scratching standardized odor-impregnated test booklets. Four booklets with 10 questions in each booklet on odor identification. Patients were asked to identify the odor by scratching the test area then selecting their answer using multiple-choice format that lists 4 different possible answers for each question. The mean change in the UPSIT was determined by comparing the score from Week 5 to the score in Week 25. The test is a forced-choice test meaning the patient is required to mark one of the four answers even if a smell is not perceived. Scores are based on number of correctly identified odors (score range 0 to 40). Higher scores indicate subject's ability to correctly identify odors.
  Reported data is a difference in the UPSIT score between Week 25 and Week 5.
Time Frame: Week 5 and Week 25
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
score on a scale | 6.6 (2.2) | 4.3 (2.5)

5. Secondary Outcome: Change in Absolute Eosinophil Count
Description: Complete Blood Count (CBC) to determine change in absolute eosinophil count. Normal Range 30-300 cells/uL.
Time Frame: Assessed at Treatment Week 0 and Week 20
Measure: Mean (Standard Error); unit: cells/uL
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
cells/uL | 678 (119) | 196.7 (171)

6. Secondary Outcome: Utilization of Prednisone as a Rescue Medication
Description: Use of Prednisone as a rescue medication during the treatment phase (week 0 through week 20) was measured in total milligrams (mg) that were taken by participant.
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
mg | 302.5 (407.77) | 297.5 (294.12)

7. Secondary Outcome: Time to Surgery
Time Frame: 24 weeks
Population: Time to nasal polyp surgery post treatment was not assessed and no data was collected.
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Dropped Out
Description: Number of participants who dropped out monitored continuously throughout the study up to 29 weeks.
Time Frame: Up to 29 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab Treatment Group | Placebo Group
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 9 months (from date of signed consent to 30 days after completion of therapy).
Arm/Group | Benralizumab Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab Treatment Group (N=12) | Placebo Group (N=12)
Upper Respiratory Infection (URI) (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03450083/Prot_SAP_000.pdf